CLINICAL TRIAL: NCT03605082
Title: A Single-center, Investigator-blind, Subject Blind, Randomized, Placebo-controlled Study to Evaluate Safety and Tolerability and Pharmacokinetics of Single Doses of UCB0107 in Healthy Japanese Subjects
Brief Title: A Study to Test the Safety and Tolerability and Pharmacokinetics of Single Doses of UCB0107 in Healthy Japanese Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: UCB Biopharma S.P.R.L. (Industry)
Responsible Party: Sponsor
Organization: UCB Pharma (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: UP0065; 2018-000475-32 (EudraCT Number)
Record Dates: First submitted 2018-06-29; First posted 2018-07-30 (Actual); Last update posted 2019-03-14 (Actual); Status verified 2019-03

CONDITIONS: Healthy Japanese Volunteers
Keywords: UCB0107; Phase 1

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- UCB0107 (Experimental): Subjects will be randomized to receive a predefined dosage of UCB0107 in order to maintain the blinding.
  Interventions: Drug: UCB0107
- Placebo (Placebo Comparator): Subjects will be randomized and receive a placebo in order to maintain the blinding.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: UCB0107 — * Pharmaceutical form: solution for infusion
  * Route of administration: intravenous use
  Arms: UCB0107
Other: Placebo — * Pharmaceutical form: solution for infusion
  * Route of administration: intravenous use
  Arms: Placebo

SUMMARY:
The purpose of the study is to evaluate the safety and tolerability and serum Pharmacokinetics (PK) of single doses of UCB0107 administered in healthy Japanese subjects.

ELIGIBILITY:
Inclusion Criteria:

* Subject is male or female, >=20 and <=75 years of age
* Subject is of Japanese descent as evidenced by appearance and verbal confirmation of familial heritage (a subject has all 4 Japanese grandparents born in Japan)
* Subject has a body mass index (BMI) >=18.0 and <=30.0 kg/m^2, with a body weight of at least 50 kilogram (kg) for males and 45 kg for females, and maximum 100 kg
* Subject is in good physical and mental health, in particular is not affected by any neurological disorder, in the opinion of the Investigator, as determined on the basis of medical history and a general clinical examination at Screening
* Subject has clinical laboratory test results within the reference ranges of the laboratory
* Subject has Blood pressure and pulse rate within normal range in supine position after 5 minutes rest
* Subject's electrocardiogram (ECG) is considered "normal," or "abnormal" but clinically nonsignificant (as interpreted by the Investigator)

Exclusion Criteria:

* Subject has any clinically relevant abnormal findings in physical examination, laboratory tests, vital signs, or electrocardiogram, which, in the opinion of the Investigator, may place the subject at risk because of participation in the study
* Subject has a history of recurrent headaches, including migraine
* Subject has a history of alcohol and/or drug abuse up to 6 months before Screening
* Subject smokes on average >5 cigarettes/day (or equivalent) during the last 3 months and is not able to stop smoking during the In-Clinic Period
* Subject has any clinically relevant brain magnetic resonance imaging (MRI) abnormality at Screening
* Subject has >upper limit of normal (ULN) of any of the following: alanine aminotransferase (ALT), aspartate aminotransferase (AST), alkaline phosphatase (ALP), or total bilirubin (≥1.5xULN total bilirubin if known Gilbert's syndrome). If subject has elevations only in total bilirubin that are >ULN and <1.5xULN, fractionate bilirubin to identify possible undiagnosed Gilbert's syndrome (ie, direct bilirubin <35%)
* Subject has a lifetime history of suicide attempt (including an actual attempt, interrupted attempt, or aborted attempt), or has suicidal ideation in the past 2 years
* Subject has a positive serology test for hepatitis B surface antigen, hepatitis B core antibodies, hepatitis C virus antibodies or antibodies to human immunodeficiency virus (HIV) type 1 and/or type 2 at Screening
* Subject has a known hypersensitivity to any components of the investigational medicinal product (IMP), comparative drugs, any biologic or small molecule, or concomitant medication as stated in this protocol
* Female subject who is breastfeeding, pregnant, or plans to become pregnant during the study or within 6 months following the final dose of the IMP

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2018-07-25 (Actual); Primary Completion 2019-03-11 (Actual); Study Completion 2019-03-11 (Actual)

PRIMARY OUTCOMES:
The incidence of treatment-emergent adverse events during the study from first dose of UCB0107 to safety follow-up/withdraw | From first dose of UCB0107 to safety follow-up/withdraw on day 140 +/-4 days
  An adverse event (AE) is any untoward medical occurrence in a patient or clinical investigation subject administered a pharmaceutical product that does not necessarily have a causal relationship with this treatment.
Maximum observed serum concentration of UCB0107 during the study | The blood sampling time points for serum Pharmacokinetics will be as follows: predose (<=60 minutes before dosing); end of infusion, 4, 6, 8, 12, 24, 36, 48, 72 and 96 hours postdose; and on Day 7, 14, 28, 42, 56, 84 and 140
  Pharmacokinetic variable:
  Cmax: maximum observed serum concentration
Area under the concentration-time curve from time 0 to infinity of UCB0107 during the study | The blood samples for serum Pharmacokinetics will be taken from predose to Day 140
  Pharmacokinetic variable:
  AUC: area under the concentration-time curve from time 0 to infinity
Area under the concentration-time curve from time 0 to time t of UCB0107 during the study | The blood sampling time points for serum Pharmacokinetics will be as follows: predose (<=60 minutes before dosing); end of infusion, 4, 6, 8, 12, 24, 36, 48, 72 and 96 hours postdose; and on Day 7, 14, 28, 42, 56, 84 and 140
  Pharmacokinetic variable:
  AUC(0-t): area under the concentration-time curve from time 0 to time t, the time of the last quantifiable concentration
Terminal half-life of UCB0107 during the study | The blood sampling time points for serum Pharmacokinetics will be as follows: predose (<=60 minutes before dosing); end of infusion, 4, 6, 8, 12, 24, 36, 48, 72 and 96 hours postdose; and on Day 7, 14, 28, 42, 56, 84 and 140
  Pharmacokinetic variable:
  t1/2: terminal half-life
Volume of distribution of UCB0107 during the study | The blood sampling time points for serum Pharmacokinetics will be as follows: predose (<=60 minutes before dosing); end of infusion, 4, 6, 8, 12, 24, 36, 48, 72 and 96 hours postdose; and on Day 7, 14, 28, 42, 56, 84 and 140
  Pharmacokinetic variable:
  Vz: volume of distribution
The clearance of UCB0107 during the study | The blood sampling time points for serum Pharmacokinetics will be as follows: predose (<=60 minutes before dosing); end of infusion, 4, 6, 8, 12, 24, 36, 48, 72 and 96 hours postdose; and on Day 7, 14, 28, 42, 56, 84 and 140
  Pharmacokinetic variable:
  CL: clearance
The time to maximum observed serum concentration of UCB0107 during the study | The blood sampling time points for serum Pharmacokinetics will be as follows: predose (<=60 minutes before dosing); end of infusion, 4, 6, 8, 12, 24, 36, 48, 72 and 96 hours postdose; and on Day 7, 14, 28, 42, 56, 84 and 140
  Pharmacokinetic variable:
  tmax: time to maximum observed serum concentration

CONTACTS AND LOCATIONS:
Overall Officials: UCB Cares, Study Director — 001 844 599 2273 (UCB)
Locations (1):
- Up0065 001, London, United Kingdom